CLINICAL TRIAL: NCT02573090
Title: SEAL-DK: Sealing Manifest Occlusal Caries Lesions in the Permanent Dentition in Children and Adolescents. RCT
Brief Title: Sealing Manifest Occlusal Caries Lesions in the Permanent Dentition
Acronym: SEAL-DK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Public Dental Health Care System, Denmark (Other)
Responsible Party: Principal Investigator, Azam Bakhshandeh, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCopenhagen1
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Dental Caries
Keywords: Occlusal caries; Resin based fissure sealant; Composite resin restoration; Effectiveness; Longevity
MeSH Terms: conditions — Dental Caries | interventions — calcium sulfate, zinc oxide, vinyl acetate, zinc phosphate root canal filling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-invasive resin based fissure sealing (Experimental): Application of resin based fissure sealing after acid etching of carious occlusal surface
  Interventions: Procedure: Non-invasive resin based fissure sealing
- Invasive resin based restoration (Active Comparator): Application of resin based resin restoration after operative intervention of caries lesion, excavation and preparation on occlusal surface
  Interventions: Procedure: Invasive resin based restoration

INTERVENTIONS:
Procedure: Non-invasive resin based fissure sealing — The dentists use resin based fissure sealants of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Cariology and Endodontics, University of Copenhagen, DK
  Other Names: Sealing
  Arms: Non-invasive resin based fissure sealing
Procedure: Invasive resin based restoration — The dentists use preparation design and resin composites of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Cariology and Endodontics, University of Copenhagen, DK
  Other Names: Restoration
  Arms: Invasive resin based restoration

SUMMARY:
The research project "SEAL-DK" is focusing on advantages and disadvantages of two treatment strategies: non-invasive fissure sealing and invasive restorative treatment of manifest occlusal caries lesions in permanent teeth in children and adolescents. The purpose of the project is to promote the understanding of the possibilities of non-invasive treatment of occlusal caries lesions in the permanent dentition, and to increase the present knowledge about the optimal threshold for sealing or restoration, respectively, when treating such lesions.

The project is carried out as a randomized study of the two treatment strategies: non-invasive versus invasive treatment of occlusal caries. When organizing the study, it is emphasized that no treatment shall be carried out, if conflicting the participating dentists' perception of clinically proper caries treatment, and that the results shall have a high reliability and consistency.

The hypothesis is that caries progression can be stopped by non-invasive fissure sealing changing the threshold and postponing the time for invasive restoration.

DETAILED DESCRIPTION:
Background: The first restoration is fatal for the prognosis of the tooth. Studies have shown that caries progression can be stopped with a tight sealing which may even lead to re-mineralization of lesions.

Aim: To investigate the possibility of treating manifest occlusal caries with non-invasive sealing instead of conventional resin restoration.

Study design: the study is carried out as a prospective, randomized clinical study (RCT). Primary, occlusal caries lesions in 521 patients, aged 6-17 years old were treated by non-invasive resin based sealing (n= 368) or resin based restoration (n=153). The dentists or patients were not free to choose the treatment type. Randomization between sealing and restoration (2:1) was made by computer for each practitioner at the University of Copenhagen and kept at the clinics in sealed envelopes. The treatments are examined clinically and radiographically after 1, 2, 3, 5, 7 and 10 years. The treatments are performed and controlled by 68 general practitioners from Public Dental Health Care Service in 9 Danish municipalities.

Sealing: The dentists use material of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Cariology and Endodontics, University of Copenhagen.

Restoration: The dentists use preparation design and material of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Cariology and Endodontics, University of Copenhagen.

The prevalence of regression, arrest and progression of sealed and restored caries lesions, are computed and related to the clinical and radiological registrations of patient, dentist or treatment related factors for assessing of statistically significant correlations.

The influence of each factor on the quality, longevity and need for retreatment of occlusal sealants and restorations, will be assessed using non-parametric tests and Kaplan-Meier survival analyses for statistical treatment of data, supplemented with summarizing multivariate survival analyses such as the Cox regression model and discriminatory analyses.

ELIGIBILITY:
Inclusion Criteria:

* each patient should have one manifest occlusal caries lesion in need of restorative treatment
* the radiographic depth of the lesion should be limited to half through the dentin
* written informed consent from children and parents should be obtained before treatment

Exclusion Criteria:

* when the occlusal lesion had communication with an approximal caries lesion or occlusal/approximal restoration
* the tooth was hypomineralized
* in case of serious chronic diseases affecting the caries experience and activity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 521 (Actual)
Dates: Start 2006-11; Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of fissure sealants | 10 years
  Radiographical scoring system:
  1) Regression in depth of lesion (success) 2: Unchanged depth of lesion (success) 3: Progression in depth of lesion (failure)
Longevity of fissure sealants | 10 years
  Clinical scoring system:
  1) Intact sealing without caries progression (success) 2: Loss of sealant with or without caries progression (failure)

SECONDARY OUTCOMES:
Effectiveness of resin based restoration | 10 years
  Radiographical scoring system:
  1) Unchanged depth of lesion (success) 2: Progression in depth of lesion (failure)
Longevity of resin based restoration | 10
  Clinical scoring system:
  1) Intact restoration without caries progression (success) 2: Defect restoration with or without caries progression (failure)